CLINICAL TRIAL: NCT01154036
Title: A Randomized, Double-Blind, Active-Controlled, Multicenter Study of Patients With Primary Hypercholesterolemia and High Cardiovascular Risk Who Are Not Adequately Controlled With Atorvastatin 10 mg: A Comparison of the Efficacy and Safety of Switching to Coadministration Ezetimibe and Atorvastatin Versus Doubling the Dose of Atorvastatin or Switching to Rosuvastatin
Brief Title: MK0653C in High Cardiovascular Risk Patients With High Cholesterol (Switch Study)(MK-0653C-162)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653C-162; 2010_517 (Other: Merck Study Number)
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2014-02-12 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Phase I: ezetimibe (EZ) 10 mg + atorvastatin (Atorva) 10 mg (Experimental): Co-administration of EZ 10 mg tablet + Atorva 10 mg tablet; once daily for 6 weeks
  Interventions: Drug: ezetimibe 10 mg; Drug: atorvastatin
- Phase I: Atorvastatin 20 mg (Active Comparator): Atorvastatin 20 mg tablet once daily for 6 weeks
  Interventions: Drug: atorvastatin
- Phase I: Rosuvastatin 10 mg (Active Comparator): Rosuvastatin 10 mg tablet once daily for 6 weeks
  Interventions: Drug: Comparator: rosuvastatin
- Phase II: EZ 10mg+Atorva 10mg (Experimental): Participants who had previously received EZ 10 mg + Atorva 10 mg in Phase I and continued on EZ 10 mg + Atorva 10 mg once daily for 6 weeks during Phase II regardless of whether or not LDL-C goals were achieved in Phase I
  Interventions: Drug: ezetimibe 10 mg; Drug: atorvastatin
- Phase II: EZ 10mg + Atorva 20mg [A] (Experimental): Participants who had previously received Atorva 20 mg in Phase I and did not reach LDL-C goal and were switched to EZ 10 mg + Atorva 20 mg once daily for 6 weeks in Phase II
  Interventions: Drug: ezetimibe 10 mg; Drug: atorvastatin
- Phase II: Atorva 40mg (Active Comparator): Participants who had previously received Atorva 20 mg in Phase I and did not reach LDL-C goal and were switched Atorva 40 mg once daily for 6 weeks in Phase II
  Interventions: Drug: atorvastatin
- Phase II: EZ 10mg + Atorva 20mg [R] (Experimental): Participants who had previously received Rosuvastatin 10 mg in Phase I and did not reach LDL-C goal and received EZ 10 mg + Atorva 20 mg once daily for 6 weeks in Phase II
  Interventions: Drug: ezetimibe 10 mg; Drug: atorvastatin
- Phase II: Rosuvastatin 20mg (Active Comparator): Participants who had previously received Rosuvastatin 10 mg in Phase I and did not reach LDL-C goal and were switched to Rosuvastatin 20 mg once daily for 6 weeks in Phase
  Interventions: Drug: Comparator: rosuvastatin

INTERVENTIONS:
Drug: ezetimibe 10 mg
  Arms: Phase I: ezetimibe (EZ) 10 mg + atorvastatin (Atorva) 10 mg; Phase II: EZ 10mg + Atorva 20mg [A]; Phase II: EZ 10mg + Atorva 20mg [R]; Phase II: EZ 10mg+Atorva 10mg
Drug: atorvastatin
  Arms: Phase I: Atorvastatin 20 mg; Phase I: ezetimibe (EZ) 10 mg + atorvastatin (Atorva) 10 mg; Phase II: Atorva 40mg; Phase II: EZ 10mg + Atorva 20mg [A]; Phase II: EZ 10mg + Atorva 20mg [R]; Phase II: EZ 10mg+Atorva 10mg
Drug: Comparator: rosuvastatin
  Arms: Phase I: Rosuvastatin 10 mg; Phase II: Rosuvastatin 20mg

SUMMARY:
This study will compare the lipid-altering efficacy and safety of switching to co-administration of ezetimibe and atorvastatin versus treatment with atorvastatin or rosuvastatin in high cardiovascular risk patients with hypercholesterolemia who have not achieved specified low-density lipoprotein cholesterol (LDL-C) levels. The primary hypothesis is that the co-administration of ezetimibe 10 mg and atorvastatin 10 mg will be superior to both atorvastatin 20 mg and rosuvastatin 10 mg with respect to the percentage reduction in low-density lipoprotein-cholesterol (LDL-C) after 6 weeks of treatment.

DETAILED DESCRIPTION:
This is a 18 week randomized, double-blind, active-controlled, multicenter study composed of a 6 week screening/run-in and 12 week double-blind treatment period (composed of 2 phases; each 6 weeks in duration). Only those participants who do not meet low density lipoprotein-cholesterol (LDL-C) goals at the end of Phase I (Week 6), were eligible to continue into Phase II (Week 12).

ELIGIBILITY:
Inclusion Criteria:

* Patient is at high cardiovascular risk and meets one of the following conditions: has never taken lipid-lowering therapy or has been off such therapy for at least 6 weeks; or, is currently taking a stable dose of certain lipid-lowering agents
* Patient is willing to maintain a cholesterol lowering diet during the study
* Female patients receiving non-cyclical hormone therapy have maintained a stable dose and regimen for at least 8 weeks and are willing to continue the same regimen during the study

Exclusion Criteria:

* Patient is Asian
* Patient routinely has more than 2 alcoholic drinks per day
* Female patient is pregnant or breastfeeding
* Patient has congestive heart failure
* Patient has had a myocardial infarction, coronary bypass surgery, angioplasty, or acute coronary syndrome within 3 months of screening
* Patient has uncontrolled cardiac arrhythmias
* Patient has had a partial ileal or gastric bypass or other significant intestinal malabsorption
* Patient has uncontrolled high blood pressure
* Patient has kidney disease
* Patient has any disease known to influence blood lipid levels
* Patient has any disorders of the blood, digestive system, or nervous system including stroke and degenerative disease that would limit study participation
* Patient has poorly controlled or newly diagnosed diabetes
* Patient is known to be HIV positive
* Patient has a history of cancer in the last 5 years, except certain skin and cervical cancers

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1547 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Krempf M, Simpson RJ Jr, Ramey DR, Brudi P, Giezek H, Tomassini JE, Lee R, Farnier M. Patient and physician factors influence decision-making in hypercholesterolemia: a questionnaire-based survey. Lipids Health Dis. 2015 May 19;14:45. doi: 10.1186/s12944-015-0037-y. PMID 25985907
- [Derived] Bays HE, Averna M, Majul C, Muller-Wieland D, De Pellegrin A, Giezek H, Lee R, Lowe RS, Brudi P, Triscari J, Farnier M. Efficacy and safety of ezetimibe added to atorvastatin versus atorvastatin uptitration or switching to rosuvastatin in patients with primary hypercholesterolemia. Am J Cardiol. 2013 Dec 15;112(12):1885-95. doi: 10.1016/j.amjcard.2013.08.031. Epub 2013 Sep 21. PMID 24063830

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in the Atorvastatin 20mg and Rosuvastatin 10mg arms who did not meet low density lipoprotein-cholesterol goals during Phase I were eligible for Phase II. Approximately 25% of participants in the ezetimibe 10mg+atorvastatin10mg arm continued to Phase II regardless of LDL-C control but were not included in any of the statistical analyses
Groups:
- Phase I: Rosuvastatin 10 mg: Rosuvastatin 10 mg tablet once daily for 6 weeks;
- Phase II: Rosuvastatin 20mg: Participants who had previously received Rosuvastatin 10 mg in Phase I and did not reach LDL-C goal and were switched to Rosuvastatin 20 mg once daily for 6 weeks in Phase II
Period: Phase I
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Phase I: Rosuvastatin 10 mg | Phase II: EZ 10mg+Atorva 10mg | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg
Started | 120 | 483 | 944 | 0 | 0 | 0 | 0 | 0
Completed | 117 (Not all completers were eligible for Phase II) | 455 (Not all completers were eligible for Phase II) | 888 (Not all completers were eligible for Phase II) | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 28 | 56 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 6 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 3 | 9 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 10 | 29 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 11 | 12 | 0 | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Phase I: Rosuvastatin 10 mg | Phase II: EZ 10mg+Atorva 10mg | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg
Started | 0 | 0 | 0 | 28 (Only participants who did not meet LDL-C goals at the end of Phase I, were eligible for Phase II) | 124 (Only participants who did not meet LDL-C goals at the end of Phase I, were eligible for Phase II) | 126 (Only participants who did not meet LDL-C goals at the end of Phase I, were eligible for Phase II) | 234 (Only participants who did not meet LDL-C goals at the end of Phase I, were eligible for Phase II) | 206 (Only participants who did not meet LDL-C goals at the end of Phase I, were eligible for Phase II)
Completed | 0 | 0 | 0 | 27 | 116 | 121 | 225 | 200
Not Completed | 0 | 0 | 0 | 1 | 8 | 5 | 9 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 4 | 2 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Phase I: Rosuvastatin 10 mg | Total
Number analyzed (Participants) | 120 | 483 | 944 | 1547
Age, Customized [Number; unit: Participants]
  <20 years | 0 | 0 | 1 | 1
  20 to 29 years | 0 | 4 | 2 | 6
  30 to 39 years | 1 | 13 | 25 | 39
  40 to 49 years | 16 | 50 | 99 | 165
  50 to 59 years | 37 | 170 | 324 | 531
  60 to 64 years | 27 | 87 | 183 | 297
  ≥65 years | 39 | 159 | 310 | 508
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 253 | 489 | 813
  Male | 49 | 230 | 455 | 734

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein-Cholesterol (LDL-C) (Phase I)
Description: LDL-C levels measured at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4. LDL-C was calculated using the Friedewald method when triglyceride (TG)<350 mg/dL (3.95 mmol/L) and beta quantification ultracentrifugation when TG≥350 mg/dL (3.95 mmol/L).
Time Frame: Baseline and Week 6 (end of Phase I )
Population: Efficacy analyses were performed using the Full Analysis Set (FAS). For Phase I this population consisted of all randomized participant who received at least one dose of study drug during Phase I and had a baseline or at least one measurement available during Phase I
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Phase I: Rosuvastatin 10 mg
Number analyzed (Participants) | 120 | 480 | 939
Percentage Change | -24.8 (23.6) | -10.1 (20.8) | -13.8 (22.8)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression — The primary hypotheses were tested at 0.045, applying Hochberg's procedure; M-Estimates, 95% CI, and p-value obtained from a robust regression model with terms for treatment and baseline values, after imputing missing values; Difference in M-estimates = -12.7, 95% CI 2-sided [-16.6 to -8.7]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Rosuvastatin 10 mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression — The primary hypotheses were tested at 0.045, applying Hochberg's procedure; [statistical method as in outcome 1, analysis 1]; Difference in M-estimate = -9.1, 95% CI 2-sided [-12.9 to -5.4]

2. Secondary Outcome: Percent Change From Baseline in Low-Density Lipoprotein-Cholesterol (LDL-C) (Phase II).
Description: LDL-C levels measured at Baseline (Week 6; end of Phase 1) and after 6 weeks of study drug administration (Week 12). Baseline was defined as the average of the values at Visits 5 and 6. LDL-C was calculated using the Friedewald method when triglyceride (TG)<350 mg/dL (3.95 mmol/L) and beta quantification ultracentrifugation when TG ≥350 mg/dL (3.95 mmol/L).
Time Frame: Baseline (Week 6) and Week 12
Population: Full Analysis Set (FAS). For Phase II this population consisted of all randomized participants who completed Phase I and were not adequately controlled at the end of Phase I, received at least 1 dose of study treatment during Phase II, had a baseline measurement for Phase II or had at least 1 measurement after the start of Phase II
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 124 | 124 | 231 | 205 | 28
Percentage Change | -16.4 (31.1) | -8.1 (23.3) | -19.3 (32.1) | -8.4 (20.8) | 2.4 (27.4)
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression — The secondary hypotheses were tested at an adaptive alpha level depending on the hypotheses testing result of the primary hypotheses; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -10.5, 95% CI 2-sided [-15.9 to -5.1]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -9.5, 95% CI 2-sided [-13.6 to -5.5]

3. Secondary Outcome: Percentage of Participants That Reach Target LDL-C Level of < 100 mg/dL (Phase I)
Time Frame: Week 6 (End of Phase I)
Population: Efficacy analyses were performed using the Full Analysis Set (FAS). For Phase I this population consisted of all randomized participants who received at least 1 dose of study drug during Phase I, had a baseline measurement for Phase I and had at least 1 measurement after the start of study drug provided during Phase I.
Measure: Number; unit: Percentage of Participants
Groups:
- Rosuvastatin 10 mg: Rosuvastatin 10 mg tablet once daily for 6 weeks;
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Rosuvastatin 10 mg
Number analyzed (Participants) | 119 | 471 | 915
Percentage of Participants | 56.3 (4.55) | 37.4 (2.23) | 43.6 (1.64)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression Model; Logistic regression model included terms for treatment and baseline LDL-C (where baseline LDL-C was fitted as 3 categories based on tertiles); Odds Ratio (OR) = 2.51, 95% CI 2-sided [1.62 to 3.89]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Rosuvastatin 10 mg; Test type: Superiority or Other; p = 0.007, Logistic Regression Model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.17 to 2.67]

4. Secondary Outcome: Percentage of Participants That Reach Target LDL-C Level of < 100 mg/dL (Phase II)
Time Frame: Week 12 (End of Phase II)
Population: Full Analysis Set (FAS). For Phase II this population consisted of all randomized participants who completed Phase I and were not adequately controlled at the end of Phase I, received at least 1 dose of study treatment during Phase II, had a baseline measurement for Phase II and had at least 1 measurement after the start of Phase II
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 120 | 123 | 228 | 201 | 28
Percentage of Participants | 55.8 (4.53) | 34.1 (4.28) | 53.5 (3.30) | 35.8 (3.38) | NA — Study plan did not include the collection of data for this arm for this Phase II endpoint; data not obtained or recorded
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p < 0.001, Logistic regression Model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 2.71, 95% CI 2-sided [1.55 to 4.73]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p < 0.001, Logistic Regression Model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 2.38, 95% CI 2-sided [1.56 to 3.63]

5. Secondary Outcome: Percentage of Participants That Reach Target LDL-C Level of < 70 mg/dL (Phase I)
Time Frame: Week 6 (End of Phase I)
Population: as for outcome 3
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Rosuvastatin 10 mg
Number analyzed (Participants) | 119 | 471 | 915
Percentage of Participants | 19.3 (3.62) | 3.0 (0.78) | 6.6 (0.82)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression Model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 9.46, 95% CI 2-sided [4.56 to 19.62]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Rosuvastatin 10 mg; Test type: Superiority or Other; p < 0.001, Logistic Regression Model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 3.90, 95% CI 2-sided [2.23 to 6.82]

6. Secondary Outcome: Percentage of Participants That Reach Target LDL-C Level of < 70 mg/dL (Phase II)
Time Frame: Week 12 (end of Phase II)
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 120 | 123 | 228 | 201 | 28
Percentage of Participants | 18.3 (3.53) | 0.8 (0.81) | 15.4 (2.39) | 3.0 (1.20) | NA — Study plan did not include the collection of data for this arm for this Phase II endpoint; data not obtained or recorded
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p = 0.001, Logistic Regression Model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 27.77, 95% CI 2-sided [3.64 to 211.83]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p < 0.001, Logistic Regression Model; [statistical method as in outcome 3, analysis 1]; Odds Ratio (OR) = 7.08, 95% CI 2-sided [2.85 to 17.56]

7. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) (Phase I)
Description: TC measured at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4
Time Frame: Baseline and Week 6 (end of Phase I)
Population: Efficacy analyses were performed using the Full Analysis Set (FAS). For Phase I this population consisted of all randomized participants who received at least 1 dose of study drug during Phase I, had a baseline measurement for Phase I or had at least 1 measurement after the start of study drug provided during Phase I.
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Rosuvastatin 10 mg
Number analyzed (Participants) | 120 | 480 | 939
Percentage Change | -13.6 (17.0) | -6.3 (14.1) | -8.2 (14.7)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -7.1, 95% CI 2-sided [-9.7 to -4.4]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Rosuvastatin 10 mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -5.8, 95% CI 2-sided [-8.3 to -3.3]

8. Secondary Outcome: Percent Change From Baseline in Total Cholesterol (TC) (Phase II)
Description: TC levels measured at Baseline (end of Phase 1) and after 6 weeks of study drug administration (Week 12; end of Phase II). Baseline was defined as the average of the values at Visits 5 and 6.
Time Frame: Baseline (Week 6; end of Phase I) and Week 12 (end of Phase II)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 124 | 124 | 231 | 205 | 28
Percentage Change | -10.2 (19.9) | -2.9 (15.7) | -13.1 (22.8) | -5.0 (14.0) | 2.2 (15.4)
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -6.8, 95% CI 2-sided [-10.7 to -3.0]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -7.4, 95% CI 2-sided [-10.2 to -4.5]

9. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG) (Phase I)
Description: TG measured at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4. Baseline and post-baseline measurements were log-transformed in the response vector, with fixed effects for treatment, time and the interaction of time by treatment.
Time Frame: Baseline and Week 6 (end of Phase I)
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Rosuvastatin 10 mg
Number analyzed (Participants) | 119 | 471 | 915
Percentage Change | -6.0 [-10.9 to -0.8] | -3.9 [-6.5 to -1.2] | -1.1 [-3.1 to 0.9]
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p = 0.466, Constrained Longitudinal Data Analysis; Geometric mean percent changes from baseline were calculated based on back-transformation via exponentiation of the model-based least square means; Difference in least-squares means = -2.1, 95% CI 2-sided [-7.8 to 3.5]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Rosuvastatin 10 mg; Test type: Superiority or Other; p = 0.081, Constrained Longitudinal Analysis; [statistical method as in outcome 9, analysis 1]; Difference in Least-squares means = -4.9, 95% CI 2-sided [-10.3 to 0.5]

10. Secondary Outcome: Percent Change From Baseline in Triglycerides (TG) (Phase II)
Description: TG levels measured at Baseline (Week 6: end of Phase I) and after 6 weeks of study drug administration (Week 12; end of Phase II). Baseline was defined as the average of the values at Visits 5 and 6. Baseline and post-baseline measurements were log-transformed in the response vector, with fixed effects for treatment, time and the interaction of time by treatment.
Time Frame: Baseline (Week 6; end of Phase I) and Week 12 (end of Phase II)
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 120 | 123 | 228 | 201 | 28
Percentage Change | -5.9 [-11.0 to -0.4] | -3.1 [-8.4 to 2.4] | -10.2 [-13.9 to -6.4] | -3.2 [-7.3 to 1.2] | NA [NA to NA] — Study plan did not include the calculation of these values
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p = 0.466, Constrained Longitudinal Data Analysis; [statistical method as in outcome 9, analysis 1]; Difference in Least-squares Means = -2.8, 95% CI 2-sided [-10.2 to 4.7]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p = 0.011, Constrained Longitudinal Data Analysis; [statistical method as in outcome 9, analysis 1]; Difference in Least-squarres Means = -7.1, 95% CI 2-sided [-12.6 to -1.6]

11. Secondary Outcome: Percent Change From Baseline in High-density Lipoprotein-Cholesterol (HDL-C) (Phase I)
Description: HDL-C measured at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4
Time Frame: Baseline and Week 6 (end of Phase I)
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Rosuvastatin 10 mg
Number analyzed (Participants) | 120 | 480 | 939
Percentage Change | 0.9 (11.9) | -1.3 (11.6) | 1.0 (13.1)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p = 0.133, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M--estimates = 1.7, 95% CI 2-sided [-0.5 to 4.0]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Rosuvastatin 10 mg; Test type: Superiority or Other; p = 0.610, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -0.6, 95% CI 2-sided [-2.7 to 1.6]

12. Secondary Outcome: Percent Change From Baseline in HDL-C (Phase II)
Description: HDL-C levels measured at Baseline (end of Phase 1) and after 6 weeks of study drug administration (Week 12; end of Phase II). Baseline was defined as the average of the values at Visits 5 and 6.
Time Frame: Baseline (Week 6; end of Phase I) and Week 12 (end of Phase II)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 124 | 124 | 231 | 205 | 28
Percentage Change | 0.9 (14.1) | 1.0 (16.0) | -0.8 (13.7) | 0.0 (15.2) | 0.0 (11.7)
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p = 0.520, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -1.0, 95% CI 2-sided [-4.2 to 2.1]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p = 0.567, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -0.7, 95% CI 2-sided [-3.1 to 1.7]

13. Secondary Outcome: Percent Change From Baseline in Apolipoprotein B (Apo B) (Phase I)
Description: Apo-B measured at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4
Time Frame: Baseline and Week 6 (end of Phase I)
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Rosuvastatin 10 mg
Number analyzed (Participants) | 120 | 479 | 938
Percentage Change | -12.1 (20.7) | -6.1 (20.7) | -7.6 (20.1)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p = 0.003, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -5.3, 95% CI 2-sided [-8.8 to -1.8]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Rosuvastatin 10 mg; Test type: Superiority or Other; p = 0.011, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -4.3, 95% CI 2-sided [-7.7 to -1.0]

14. Secondary Outcome: Percent Change From Baseline in Apo B (Phase II)
Description: Apo-B levels measured at Baseline (Week 6; end of Phase 1) and after 6 weeks of study drug administration (Week 12; end of Phase II). Baseline was defined as the average of the values at Visits 5 and 6.
Time Frame: Baseline (Week 6; end of Phase 1) and Week 12 (end of Phase II)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 124 | 124 | 231 | 205 | 27
Percentage Change | -12.0 (26.5) | -6.3 (19.6) | -14.0 (25.1) | -4.9 (21.8) | -4.0 (16.8)
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p = 0.079, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -4.3, 95% CI 2-sided [-9.2 to 0.5]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -7.7, 95% CI 2-sided [-11.4 to -4.1]

15. Secondary Outcome: Percent Change From Baseline in Apolipoprotein A-I (Apo A-I) (Phase I)
Description: Apo-A-I measured at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4
Time Frame: Baseline and Week 6 (end of Phase I)
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Rosuvastatin 10 mg
Number analyzed (Participants) | 120 | 479 | 938
Percentage Change | -0.6 (13.1) | -1.9 (12.5) | 1.4 (13.0)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p = 0.156, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = 1.6, 95% CI 2-sided [-0.6 to 3.8]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Rosuvastatin 10 mg; Test type: Superiority or Other; p = 0.425, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -0.9, 95% CI 2-sided [-2.9 to 1.2]

16. Secondary Outcome: Percent Change From Baseline in Apo A-I (Phase II)
Description: Apo-A-I levels measured at Baseline (end of Phase 1) and after 6 weeks of study drug administration (Week 12; end of Phase II). Baseline was defined as the average of the values at Visits 5 and 6.
Time Frame: Baseline (Week 6; end of Phase I) and Week 12 (end of Phase II)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 124 | 124 | 231 | 205 | 27
Percentage Change | 1.6 (11.9) | 1.4 (14.1) | -0.6 (14.4) | 0.0 (16.0) | -0.7 (14.3)
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p = 0.739, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = 0.5, 95% CI 2-sided [-2.5 to 3.6]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p = 0.410, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -1.0, 95% CI 2-sided [-3.3 to 1.3]

17. Secondary Outcome: Percent Change From Baseline in Non-HDL-C (Phase I)
Description: Non-HDL-C measured at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4
Time Frame: Baseline and Week 6 (end of Phase I)
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Rosuvastatin 10 mg
Number analyzed (Participants) | 120 | 480 | 939
Percentage Change | -18.0 (22.3) | -7.9 (17.6) | -11.1 (19.8)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -10.1, 95% CI 2-sided [-13.6 to -6.6]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Rosuvastatin 10 mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -7.6, 95% CI 2-sided [-10.9 to -4.3]

18. Secondary Outcome: Percent Change From Baseline in Non-HDL-C (Phase II)
Description: Non-HDL-C levels calculated at Baseline (end of Phase 1) and after 6 weeks of study drug administration (Week 12; end of Phase II). Baseline was defined as the average of the values at Visits 5 and 6.
Time Frame: Baseline (Week 6; end of Phase I) and Week 12 (end of Phase II)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 124 | 124 | 231 | 205 | 28
Percentage Change | -17.5 (26.1) | -5.5 (16.6) | -18.1 (29.4) | -6.3 (18.5) | -0.5 (17.7)
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -9.3, 95% CI 2-sided [-14.0 to -4.5]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p = 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -9.8, 95% CI 2-sided [-13.5 to -6.2]

19. Secondary Outcome: Percent Change From Baseline in TC/HDL-C Ratio (Phase I)
Description: TC/HDL-C ratio calculated at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4
Time Frame: Baseline and Week 6 (end of Phase I)
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Rosuvastatin 10 mg
Number analyzed (Participants) | 120 | 480 | 939
Percentage Change | -14.3 (17.9) | -4.5 (16.8) | -9.0 (19.1)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -8.1, 95% CI 2-sided [-11.2 to -4.9]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Rosuvastatin 10 mg; Test type: Superiority or Other; p = 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -4.8, 95% CI 2-sided [-7.8 to -1.9]

20. Secondary Outcome: Percent Change From Baseline in TC/HDL-C Ratio (Phase II)
Description: TC/HDL-C Ratio calculated at Baseline (end of Phase 1) and after 6 weeks of study drug administration (Week 12; end of Phase II). Baseline was defined as the average of the values at Visits 5 and 6.
Time Frame: Baseline (Week 6; end of Phase 1) and Week 12 (end of Phase II)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 124 | 124 | 231 | 205 | 28
Percentage Change | -13.5 (21.7) | -6.5 (13.9) | -11.7 (23.3) | -4.0 (17.8) | -1.0 (9.6)
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -6.9, 95% CI 2-sided [-11.0 to -2.8]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -6.4, 95% CI 2-sided [-9.4 to -3.3]

21. Secondary Outcome: Percent Change From Baseline in LDL-C/HDL-C Ratio (Phase I)
Description: LDL-C/HDL-C ratio calculated at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4
Time Frame: Baseline and Week 6 (end of Phase I)
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: Percentage Change
Groups:
- Phase 1: Rosuvastatin 10 mg: Rosuvastatin 10 mg tablet once daily for 6 weeks;
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Phase 1: Rosuvastatin 10 mg
Number analyzed (Participants) | 120 | 480 | 939
Percentage Change | -23.9 (23.6) | -7.1 (23.2) | -14.7 (26.9)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -13.7, 95% CI 2-sided [-18.1 to -9.3]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase 1: Rosuvastatin 10 mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -7.8, 95% CI 2-sided [-11.9 to -3.6]

22. Secondary Outcome: Percent Change From Baseline in LDL-C/HDL-C Ratio (Phase II)
Description: LDL-C/HDL-C Ratio calculated at Baseline (end of Phase 1) and after 6 weeks of study drug administration (Week 12; end of Phase II). Baseline was defined as the average of the values at Visits 5 and 6.
Time Frame: Baseline (Week 6; end of Phase 1) and Week 12 (end of Phase II)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 124 | 124 | 231 | 205 | 28
Percentage Change | -20.6 (31.4) | -8.2 (20.6) | -18.2 (31.6) | -7.5 (21.5) | -4.5 (22.9)
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -10.4, 95% CI 2-sided [-15.8 to -4.9]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -8.3, 95% CI 2-sided [-12.5 to -4.2]

23. Secondary Outcome: Percent Change From Baseline in Apo B/Apo A-I Ratio (Phase I)
Description: Apo B/Apo A-I ratio calculated at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4
Time Frame: Baseline and Week 6 (end of Phase I)
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Phase 1: Rosuvastatin 10 mg
Number analyzed (Participants) | 120 | 479 | 938
Percentage Change | -13.0 (22.3) | -4.8 (18.9) | -8.8 (23.0)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -6.3, 95% CI 2-sided [-10.0 to -2.5]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase 1: Rosuvastatin 10 mg; Test type: Superiority or Other; p = 0.052, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -3.5, 95% CI 2-sided [-7.1 to 0.0]

24. Secondary Outcome: Percent Change From Baseline in Apo B/Apo A-I Ratio (Phase II)
Description: Apo B/Apo A-I Ratio calculated at Baseline (Week 6; end of Phase 1) and after 6 weeks of study drug administration (Week 12; end of Phase II). Baseline was defined as the average of the values at Visits 5 and 6.
Time Frame: Baseline (Week 6; end of Phase 1) and Week 12 (end of Phase II)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 124 | 124 | 231 | 205 | 27
Percentage Change | -11.2 (26.2) | -6.4 (19.4) | -11.2 (27.5) | -5.4 (21.5) | -6.7 (11.3)
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p = 0.024, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -5.8, 95% CI 2-sided [-10.8 to -0.8]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p = 0.002, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -6.1, 95% CI 2-sided [-9.9 to -2.3]

25. Secondary Outcome: Percent Change From Baseline in Non-HDL-C/HDL-C Ratio (Phase I)
Description: Non HDL-C/HDL-C ratio calculated at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4
Time Frame: Baseline and Week 6 (end of Phase I)
Population: as for outcome 7
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Phase 1: Rosuvastatin 10 mg
Number analyzed (Participants) | 120 | 480 | 939
Percentage Change | -18.9 (23.9) | -6.3 (22.8) | -12.2 (25.9)
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -10.6, 95% CI 2-sided [-14.9 to -6.4]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase 1: Rosuvastatin 10 mg; Test type: Superiority or Other; p = 0.002, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -6.2, 95% CI 2-sided [-10.2 to -2.2]

26. Secondary Outcome: Percent Change From Baseline in Non-HDL-C/HDL-C Ratio (Phase II)
Description: Non HDL-C/HDL-C Ratio calculated at baseline (Week 6; end of Phase 1) and after 6 weeks of study drug administration (Week 12; end of Phase II). Baseline was defined as the average of the values at Visits 5 and 6.
Time Frame: Baseline (Week 6; end of Phase 1) and Week 12 (end of Phase II)
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 124 | 124 | 231 | 205 | 28
Percentage Change | -18.2 (29.5) | -8.8 (18.8) | -16.3 (32.3) | -5.9 (23.4) | -1.9 (12.9)
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -9.3, 95% CI 2-sided [-14.8 to -3.9]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p < 0.001, Multiple Imputation Robust Regression; [statistical method as in outcome 1, analysis 1]; Difference in M-estimates = -8.4, 95% CI 2-sided [-12.6 to -4.2]

27. Secondary Outcome: Percent Change From Baseline in High-sensitivity C-reactive Protein (Hs-CRP) (Phase I)
Description: hs-CRP measured at Baseline and after 6 weeks of treatment (Week 6; end of Phase I). Baseline was defined as the average value of the measurements taken at Visits 3 and 4. Baseline and post-baseline measurements were log-transformed in the response vector, with fixed effects for treatment, time and the interaction of time by treatment.
Time Frame: Baseline and Week 6 (end of Phase I)
Population: as for outcome 3
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Phase I: Rosuvastatin 10 mg
Number analyzed (Participants) | 117 | 458 | 899
Percentage Change | -10.5 [-23.0 to 4.0] | -6.6 [-13.6 to 1.0] | -9.0 [-14.0 to -3.6]
Statistical Analysis 1: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Atorvastatin 20 mg; Test type: Superiority or Other; p = 0.613, Constrained Longitudinal Data Analysis; [statistical method as in outcome 9, analysis 1]; Difference in Least-squares Means = -3.9, 95% CI 2-sided [-18.9 to 11.1]
Statistical Analysis 2: Comparison: Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg vs Phase I: Rosuvastatin 10 mg; Test type: Superiority or Other; p = 0.831, Constrained Longitudinal Data Analysis; [statistical method as in outcome 9, analysis 1]; Difference in Least-squares Means = -1.5, 95% CI 2-sided [-15.7 to 12.6]

28. Secondary Outcome: Percent Change From Baseline in Hs-CRP (Phase II)
Description: hs-CRP measured at Baseline (Week 6; end of Phase 1) and after 6 weeks of study drug administration (Week 12; end of Phase II). Baseline was defined as the average of the values at Visits 5 and 6. Baseline and post-baseline measurements were log-transformed in the response vector, with fixed effects for treatment, time and the interaction of time by treatment.
Time Frame: Baseline (Week 6; end of Phase 1) and Week 12 (end of Phase II)
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage Change
Arm/Group | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg | Phase II: EZ 10mg+Atorva 10mg
Number analyzed (Participants) | 119 | 121 | 226 | 200 | 27
Percentage Change | -19.5 [-31.5 to -5.3] | -6.4 [-20.2 to 9.8] | -10.9 [-20.9 to 0.3] | 0.7 [-11.2 to 14.2] | NA [NA to NA] — Study plan did not include the calculation of these values
Statistical Analysis 1: Comparison: Phase II: EZ 10mg + Atorva 20mg [A] vs Phase II: Atorva 40mg; Test type: Superiority or Other; p = 0.187, Constrained Longitudinal Data Analysis; [statistical method as in outcome 9, analysis 1]; Difference in Least-squares Means = -13.1, 95% CI 2-sided [-32.6 to 6.4]
Statistical Analysis 2: Comparison: Phase II: EZ 10mg + Atorva 20mg [R] vs Phase II: Rosuvastatin 20mg; Test type: Superiority or Other; p = 0.153, Constrained Longitudinal Data Analysis; [statistical method as in outcome 9, analysis 1]; Difference in Least-squares Means = -11.6, 95% CI 2-sided [-27.7 to 4.4]

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Description: Adverse events were reported using the All Patients as Treated (APaT) Population, which was defined as all randomized participants who received at least 1 dose of study drug.
Arm/Group | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg | Phase I: Atorvastatin 20 mg | Phase I: Rosuvastatin 10 mg | Phase II: EZ 10mg+Atorva 10mg | Phase II: EZ 10mg + Atorva 20mg [A] | Phase II: Atorva 40mg | Phase II: EZ 10mg + Atorva 20mg [R] | Phase II: Rosuvastatin 20mg
Serious Adverse Events (participants affected / at risk) | 0/120 | 3/480 | 10/939 | 0/28 | 2/124 | 2/124 | 5/231 | 1/205
Other Adverse Events (participants affected / at risk) | 0/120 | 0/480 | 0/939 | 0/28 | 0/124 | 0/124 | 0/231 | 0/205
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Ezetimibe (EZ) 10 mg + Atorvastatin (Atorva) 10 mg (N=120) | Phase I: Atorvastatin 20 mg (N=480) | Phase I: Rosuvastatin 10 mg (N=939) | Phase II: EZ 10mg+Atorva 10mg (N=28) | Phase II: EZ 10mg + Atorva 20mg [A] (N=124) | Phase II: Atorva 40mg (N=124) | Phase II: EZ 10mg + Atorva 20mg [R] (N=231) | Phase II: Rosuvastatin 20mg (N=205)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.